CLINICAL TRIAL: NCT06917443
Title: Abdominally Targeted Management Exercises for Crohn's Disease Patients (TAME-CD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shmuel Kivity, MD (Other Government)
Responsible Party: Sponsor-Investigator, Shmuel Kivity, MD, Professor, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0438-24-TLV; MOH_2024-11-20_013744 (Other: The Israeli ministry of health)
Record Dates: First submitted 2025-03-18; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Crohn Disease (CD); IBD (Inflammatory Bowel Disease)
Keywords: physical exercise; Crohn's disease; randomized trial
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either intervention or control arm in 2:1 ratio, respectively.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominally targeted exercises (Experimental): The interventional exercise regimen will include specific abdominally targeted exercises postulated to increase blood flow to the intestine and decrease inflammation. Patients will be asked to perform the exercises 6 days every week. Patients will be asked to complete 3 different videos repeatedly, one video per day, as many days a week as possible.
  Interventions: Other: Abdominally targeted exercises
- Generally recommended exercises (Placebo Comparator): The control arm will practice generally recommended exercises, without particular attention to the abdomen. Patients will be asked to perform the exercises 6 days every week. Patients will be asked to complete 3 different videos repeatedly, one video per day, as many days a week as possible.
  Interventions: Other: General exercises

INTERVENTIONS:
Other: Abdominally targeted exercises — The interventional exercise regimen will include specific abdominally targeted exercises postulated to increase blood flow to the intestine and decrease inflammation.
  Arms: Abdominally targeted exercises
Other: General exercises — Generally recommended exercises, without particular attention to the abdomen
  Arms: Generally recommended exercises

SUMMARY:
The goal of this clinical trial is to learn if abdominally targeted exercises can assist to manage disease activity in Crohn disease (CD) patients.

The main questions it aims to answer are:

Does abdominally targeted exercises can improve the quality of life of CD patients.

Does abdominally targeted exercises positively influence clinical and biological responses in CD patients.

Researchers will compare performing sets of special physical exercises designed for CD patients, compared to a control set of exercises ("generic" physical activity) to see if exercises designed for CD can result in an improved quality of life, in CD patients suffering from mild to moderate disease activity.

Participants will:

* Perform physical exercises designed for CD or control set of exercises every day for 8 weeks.
* Visit the clinic once every 4 weeks for doctor visit, blood and stool test and filling out questionnaires.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are chronic relapsing diseases that carry considerable impact on patients' quality of life (QoL) including objective measures such as increased bowel movements and more subjective measures such as fatigue, stress and depression. While the pathogenesis of IBD is thought to result from a deregulated immune response towards microbial antigens in a genetically predisposed person, various associations of environmental factors and disease activity have been described. These include, but are not limited to diet, stress, physical activity, and microbial composition and function.

Mild to moderate physical activity, which by itself can be beneficial for patients who suffer from chronic disabling diseases such as IBD, is thought to have positive effects on health, general well-being and stress. The positive effects of physical activity can be mediated directly and/ or secondarily through its impact on other modifying factors such as sleep quality, bowel circadian rhythm, and perceived stress. In this regard, by reducing stress through physical activity, one can not only improve patients' QoL and reported outcomes (PROMs) such as sleep quality and stress reduction, which are an important measure by themselves; but also to improve subjective measures of the disease severity. Additionally, physical activity can impact the enteric microbiome, which can be beneficial in IBD patients.

It is currently not clear whether routine physical activity, performed by IBD patients, improves their symptoms, disease activity and quality of lives and if yes, which activity is mostly recommended.

In this study, the investigator intends to further examine whether these disease-specifically designed exercise sets can improve patients' perceived QoL and positively influence clinical and biological responses.

The hypothesize anticipates performing sets of special physical exercises designed for IBD patients, compared to a control set of exercises, can result in an improved QoL, in CD patients suffering from mild to moderate disease activity.

The effect of each set of exercises on patients' QoL, clinical and biological responses through symptoms severity, inflammatory biomarkers, intestinal ultrasound, change in microbiome and gut permeability, will be evaluated.

For this aim, CD patients suffering from mild to moderate disease will be randomized to undergo either a set of specific physical exercises for CD or a control set of unrelated exercises. Patients will be randomized to either group by a computer randomization program according to disease activity (5<HBI≤7 or 7<HBI≤15) and biomarker status (Fecal calprotectin below or above 350ugr/gr). Patients will receive an email with the link to an internet site where they will be able to watch the exercise program.

Videos sets of exercises will be available online and patients will be able to watch and follow these videos at their home. Each video will include explicit instructions and examples for each of the exercises.

Compliance will be documented by the study coordinator (by mail or phone call) every week during the first 2 weeks and then every 2 weeks until the end of the study. This will be verified through the software itself, which documents whenever a patient activates the video.

All patients should remain on consistent dietary regimen throughout the study period.

Patients will attend research visits at weeks 0, 4, and 8. During visits patients will answer questionnaires for QoL (IBDQ), and PROMs (PROMIS-29); and will be monitored for disease activity. At these time points, patients will give biologic samples:

1. Serum- 20 ml of blood will be drawn for serum analysis of CRP concentration and for LPS binding protein (LBP). Serum will also be frozen for future metabolome analysis.
2. Stool - analyzed for inflammatory marker calprotectin, as well as microbial composition and function.

Data collection will include basic medical and demographic information, including gender, age, weight, height, smoking and exercise habits. Medical data will include age at diagnosis, disease duration, CD Montreal classification, HBI (Harvey-Bradshaw Index), lab results (CRP, LBP and calprotectin), comorbidities, medications history and previous intestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no treatment or on constant medicinal therapy, expected to remain constant: mesalamine for at least 6 weeks, steroids at least 2 weeks (≤20mg prednisone or budesonide ≤6mg), immunomodulatory at least 12 weeks or biologics/ small molecules for at least 12 weeks therapy. Patients who initiate the study on steroids will remain on a constant dose throughout the study.
* If patients stopped therapy prior to the study then they should be at least 2 weeks from stopping steroids or 5ASA, or 4 weeks from stopping small molecules, 8 weeks from stopping biologics, or 12 weeks from stopping thiopurines.
* CD patients will be included if their symptoms score >4 and ≤15 on the HBI score
* Fecal calprotectin>150ug/gr or evidence of an active disease per IUS defined as increased blood flow (modified Limberg score>0) or thickness of bowel wall>3mm

Exclusion Criteria:

* Inability to commit for performing at least 10-15 minutes of exercise, 6 times a week.
* Lack of availability or capability to use a computer/ internet.
* Any proven current infection such as, fever, active abscess, Clostridioides difficile infection, positive stool culture, or parasite in patients with chronic diarrhea.
* Inability to sign informed consent and/ or complete the study protocol.
* Incompetent individuals who are unable to provide informed consent.
* Planed pregnancy or pregnancy- up to 3 months post labor.
* Subjects with chronic conditions such as active arthritis, cancer (within the previous 5 years, not including BCC, SCC), organ transplant subjects, advanced kidney or liver disease, or systemic inflammatory conditions other than IBD.
* Patients who underwent surgery in the previous 3 months, had more than 1 surgery of intestinal resection, patients with ileostomy, pouch or patients with short bowel (small intestine<1.5 meter).
* Patients with a significant abdominal wall hernia, unless received a written confirmation from a treating surgeon.
* Active peri-anal disease (fistula, abscess, fissure), stricturing or penetrating disease
* Active extra-intestinal manifestations (not excluded are- oral aphthae and peripheral arthralgia without arthritis)
* Patients on total parenteral nutrition (TPN) or on exclusive enteral nutrition (EEN).
* Probiotics or antibiotics in the 15 days prior to enrollment or during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | From enrollment to the end of treatment at 8 weeks
  Clinical response rate will be assessed by using a clinical activity index, Harvey-Bradshaw index (HBI), and defined by a decrease of ≥3 points. A greater decrease is regarded as a better response.
Clinical remission rate | From enrollment to the end of treatment at 8 weeks
  Clinical remission rate will be assessed by using a clinical activity index, HBI defined by achieving HBI<5. Lower scores indicate lower disease activity and severity.
Biomarker remission rate | From enrollment to the end of treatment at 8 weeks
  biomarker remission as defined by calprotectin <150 μg/g. Lower levels indicate better outcome
Biomarker remission rate | From enrollment to the end of treatment at 8 weeks
  Biomarker remission as defined by CRP levels <5 mg/L. Lower levels indicate better outcome
Change from Baseline in mean values of PROMIS-29 scores | From enrollment to the end of treatment at 8 weeks
  To assess the differences in patients' perceived QoL according to patients reported outcomes questionnaires: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Change from Baseline in mean values of IBDQ | From enrollment to the end of treatment at 8 weeks
  To assess the differences in patients' perceived QoL according to patients reported outcomes questionnaires: Inflammatory Bowel Disease Questionnaire (IBDQ)

SECONDARY OUTCOMES:
Biomarker response rate | From enrollment to the end of treatment at 8 weeks
  Biomarker response will be assessed by a 50% decrease in fecal calprotectin. Greater decrease indicates better response.
IUS remission rate | End of treatment at 8 weeks
  IUS remission will be determined by modified Limberg score evaluating bowel wall vascularity. Score range between grade 0 to 4. Remission is defined by modified Limberg score= 0.
Clinical remission rate | From enrollment to 4 weeks
  Clinical remission rate will be assessed by using a clinical activity index, HBI defined by achieving HBI<5. Lower scores indicate lower disease activity and severity.
Clinical response rate | From enrollment to 4 weeks
  Clinical response rate will be assessed by using a clinical activity index, Harvey-Bradshaw index (HBI), and defined by a decrease of ≥3 points. A greater decrease is regarded as a better response.
Change from Baseline in mean values of PROMIS-29 scores | From enrollment to 4 weeks
  To assess the differences in patients' perceived QoL according to patients reported outcomes questionnaires: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Change from Baseline in mean values of IBDQ | From enrollment to 4 weeks
  To assess the differences in patients' perceived QoL according to patients reported outcomes questionnaires: Inflammatory Bowel Disease Questionnaire (IBDQ)

OTHER OUTCOMES:
Change from baseline in mean serum levels of LBP | From enrollment to the end of treatment at 8 weeks
  To assess LPS binding protein (LBP) serum level as a marker of permeability
Change from baseline in mean serum levels of LBP | From enrollment to 4 weeks
  To assess LPS binding protein (LBP) serum level as a marker of permeability
Treatment affect on microbiome and metabolome composition or function | From enrollment to the end of treatment at 8 weeks
  To evaluate the differences on microbiome and metabolome composition or function based on microbial metagenomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, Professor, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Department of Gastroenterology and Liver Diseases, Tel Aviv Medical Center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided